CLINICAL TRIAL: NCT06086249
Title: Clinical and Radiographic Success of Regeneration Using Injectable Platelet Rich Fibrin Versus Root Canal Treatment in Mature Permanent Molars With Apical Periodontitis: A Randomized Controlled Pilot Study
Brief Title: Clinical and Radiographic Success of Regeneration Using Injectable Platelet Rich Fibrin
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Samah Mohsen Kanzel, Pediatric Dentist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 102032
Record Dates: First submitted 2023-10-09; First posted 2023-10-17 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Apical Periodontitis
MeSH Terms: conditions — Periapical Periodontitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regeneration using Injectable platelet-rich fibrin (Experimental): A 10-mL sample of whole venous blood will be drawn from the patient's forearm (median cubital vein). It will be centrifuged immediately by a tabletop centrifuge at 700 rpm for 3 minutes at room temperature. Injectable platelet-rich fibrin (I-PRF) will be collected. After that, the I-PRF will be injected inside the canals using a plastic syringe needle that will be placed 1mm short of the working length and withdrawn gradually while injecting till reaching the orifices of the canals. After that, a Collagen membrane matrix will be placed above the canal orifice and will left for 5 minutes to partially harden, then a 3 mm thick layer of MTA will be placed directly over it. The cavity will be sealed with composite and covered with a stainless steel crown.
  Interventions: Procedure: Regeneration using Injectable platelet-rich fibrin
- Root canal treatment (Active Comparator): The root canal will be obturated with gutta-percha by the cold lateral condensation technique with epoxy resin-based root canal sealer, the cavity will be sealed with composite and covered with a stainless steel crown.
  Interventions: Procedure: Root canal treatment

INTERVENTIONS:
Procedure: Regeneration using Injectable platelet-rich fibrin — root canals of affected molars will be cleaned and shaped chemo-mechanically, after two weeks I-PRF will be applied.
  Arms: Regeneration using Injectable platelet-rich fibrin
Procedure: Root canal treatment — Conventional root canal treatment using gutta-percha obturation
  Arms: Root canal treatment

SUMMARY:
Study aimed at assessing the clinical and radiographic success of pulp regeneration using injectable platelet-rich fibrin in mature permanent molars with apical periodontitis versus root canal treatment using Gutta Percha (GP) obturation.

DETAILED DESCRIPTION:
Randomized pilot study, parallel groups design with 1:1 allocation ratio.

PICOT:

Population: Mature first permanent molar with apical periodontitis. Intervention: Regeneration using injectable platelet-rich fibrin. Control: Root canal treatment using GP obturation. outcomes: clinical and radiographic success. Source of patients: this study will be conducted in the outpatient postgraduate clinic of the Pediatric Dentistry and Dental Public Health Department - Faculty of Dentistry, Cairo University, Egypt.

Written Informed consent from participating children/parents. Baseline records photographs, clinical inspection, percussion test, periapical radiograph, and personal data collection will be conducted.

A diagnostic chart with personal, medical, and dental history will be filled Diagnosis and treatment of the cases will be performed according to the Treatment Standards of the American Association of Endodontists (AAE) 2020 of Non-Surgical Endodontics for the Uncomplicated Mature Permanent Teeth.

Allocation (concealed by withdrawing a sealed opaque envelope containing Four-folded numbered papers containing the type of treatment then writing the patient's name and I.D. on it and will be opened in the next visit).

The radiographic examination will be performed by taking a periapical X-ray using (a parallel technique) to assess the inclusion criteria. The preoperative radiograph will serve as a reference for the follow-up radiographs. Standardization of the technique to avoid any vertical dimension distortion and provide reproducible images using an X-ray holding device.

An individual XCP (Extension Cone Paralleling) index will be prepared for each patient by registering the bite to allow consistent comparisons of the radiographs.

Intra-operative procedure:

First appointment:

* Local anesthesia administration using 1.8-mL of articaine 4% with epinephrine 1:100000 using inferior alveolar nerve block.
* Rubber dam will be applied, then caries removal and access cavity preparation will be established using a sterile carbide bur no. 8, and Endo Z bur.
* Initial canal exploration will be performed with Endo Probe and no. 10 K-file to gauge canal size, shape, and configuration. Working length will be determined using an apex locator with no 15-hand K-file that will be kept 0.3 mm short of the radiographic apex and will be confirmed radiographically.
* Then, the root canal preparation will be done as follows:

Rotary instrumentation will be preceded by manual hand instrumentation using no 20 K-file to check the patency. Then, the rotary instrumentation will be done using rotary files.

EDTA gel will be used as a lubricating paste during canal preparation with rotary files.

Sodium hypochlorite (1.5%) and saline irrigation using a side vented needle into the apical third of the canal to remove debris with copious irrigation using ultrasonic irrigation.

Dryness will be done using paper points size 30. The root canal will be filled homogeneously to the working length with Calcium Hydroxide paste (Metapaste), then, a small Teflon will be applied above the orifices and the tooth will be temporarily restored with Glass Ionomer restorative material till the next appointment.

Second appointment:

All the patients will be recalled after 3 weeks, if the symptoms are suggestive of persistent infection, the root canals will be re-irrigated with sodium hypochlorite followed by saline, and reinjected with calcium hydroxide paste. If the symptoms are relieved, patients will proceed to the next step.

* A 1.8-mL of articaine 4% with epinephrine 1:100000 will be administered as inferior alveolar nerve block. The rubber dam will be placed, and the glass ionomer cement and Teflon will be removed. The root canals will be agitated with master apical K-file and re-irrigated using 17% EDTA solution followed by saline irrigation, then the canals will be dried using a paper point.
* For the intervention group, I-PRF Regeneration will be applied.
* For the control group, root canal treatment will be applied.

C) Follow up:

Clinical evaluation will be performed on 1, 3, 6, 9, and 12 months post-operatively.

Radiographic evaluation will be performed pre-operatively (baseline), and postoperative following the second appointment at 6, and 12 months using the individualized XCP (Extension Cone Paralleling) index and the Digital X-ray machine.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged between 10-15 years.
2. First Permanent molar diagnosed with apical periodontitis.
3. A cooperative and compliant patient/ parent.
4. Patients not allergic to medicaments necessary to complete the procedure.
5. Patients with no history of chronic systemic diseases.

Exclusion Criteria:

1. Teeth indicated for post and core.
2. Non-restorable tooth.
3. Previous root canal treatment.
4. Curved canal of more than 25°.
5. Periodontal pocket larger than 3 mm.
6. Teeth with developmental anomalies.

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Clinical success | 1, 3, 6, 9 and 12 months
  Clinical Success is a composite outcome and will be recorded as Clinically Successful or Clinically Unsuccessful based on the following evaluation criteria:
  Clinically Successful: Following assigned treatment in case of absence of all of the following: spontaneous pain, swelling, sinus tract, palpation pain, percussion pain.
  Clinically unsuccessful: Following assigned treatment in case of presence of any of the following: spontaneous pain, swelling, sinus tract, palpation pain, percussion pain.

SECONDARY OUTCOMES:
Radiographic success | 6 and 12 months
  The scores will be follow:
  1. Absence of the periapical lesion; if the postoperative radiographic periodontal space is smaller than 0.5 mm.
  2. Reduction of the periapical lesion; if the postoperative radiographic lesion is smaller than approximately 20% of the preoperative radiographic lesion.
  3. Enlargement of the periapical lesion; if the postoperative radiographic lesion is bigger than approximately 20% of the preoperative radiographic lesion.
  4. Uncertain: if the case cannot be defined as absence, reduction, or enlargement of the periapical lesion, periapical rarefaction 1 mm or less, extraction of tooth before recall because of reasons not related to outcome of endodontic treatment.
Overall success | 6 and 12 months
  The treatment will be scored as Success in case there is absence or reduction of the radiolucency (score 1 or 2), in addition to being clinically asymptomatic with no sinus tract, swelling, with no spontaneous, palpation, or percussions pain. On the other side, if the case showed a score of 3 or 4 radiographically or a symptomatic tooth, the case was recorded as Failure.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Youssef A, Ali M, ElBolok A, Hassan R. Regenerative endodontic procedures for the treatment of necrotic mature teeth: A preliminary randomized clinical trial. Int Endod J. 2022 Apr;55(4):334-346. doi: 10.1111/iej.13681. Epub 2022 Jan 31. PMID 35030270
- [Background] Rafiee A, Memarpour M, Najibi Y, Khalvati B, Kianpour S, Morowvat MH. Antimicrobial Efficacy of a Novel Antibiotic-Eluting Injectable Platelet-Rich Fibrin Scaffold against a Dual-Species Biofilm in an Infected Immature Root Canal Model. Biomed Res Int. 2020 Dec 8;2020:6623830. doi: 10.1155/2020/6623830. eCollection 2020. PMID 33490247
- [Background] Aydinyurt HS, Sancak T, Taskin C, Basbugan Y, Akinci L. Effects of injectable platelet-rich fibrin in experimental periodontitis in rats. Odontology. 2021 Apr;109(2):422-432. doi: 10.1007/s10266-020-00557-1. Epub 2020 Oct 17. PMID 33068206
- [Background] Taylor GD, Vernazza CR, Abdulmohsen B. Success of endodontic management of compromised first permanent molars in children: A systematic review. Int J Paediatr Dent. 2020 May;30(3):370-380. doi: 10.1111/ipd.12599. Epub 2019 Dec 13. PMID 31778237
- [Background] Nageh M, Ahmed GM, El-Baz AA. Assessment of Regaining Pulp Sensibility in Mature Necrotic Teeth Using a Modified Revascularization Technique with Platelet-rich Fibrin: A Clinical Study. J Endod. 2018 Oct;44(10):1526-1533. doi: 10.1016/j.joen.2018.06.014. Epub 2018 Aug 31. PMID 30174103
- [Background] Gollapudi M, Bajaj P, Oza RR. Injectable Platelet-Rich Fibrin - A Revolution in Periodontal Regeneration. Cureus. 2022 Aug 31;14(8):e28647. doi: 10.7759/cureus.28647. eCollection 2022 Aug. PMID 36196318
- [Background] Arslan H, Ahmed HMA, Sahin Y, Doganay Yildiz E, Gundogdu EC, Guven Y, Khalilov R. Regenerative Endodontic Procedures in Necrotic Mature Teeth with Periapical Radiolucencies: A Preliminary Randomized Clinical Study. J Endod. 2019 Jul;45(7):863-872. doi: 10.1016/j.joen.2019.04.005. Epub 2019 May 31. PMID 31155298
- [Background] Jha P, Virdi MS, Nain S. A Regenerative Approach for Root Canal Treatment of Mature Permanent Teeth: Comparative Evaluation with 18 Months Follow-up. Int J Clin Pediatr Dent. 2019 May-Jun;12(3):182-188. doi: 10.5005/jp-journals-10005-1616. PMID 31708612
- [Background] Brizuela C, Meza G, Urrejola D, Quezada MA, Concha G, Ramirez V, Angelopoulos I, Cadiz MI, Tapia-Limonchi R, Khoury M. Cell-Based Regenerative Endodontics for Treatment of Periapical Lesions: A Randomized, Controlled Phase I/II Clinical Trial. J Dent Res. 2020 May;99(5):523-529. doi: 10.1177/0022034520913242. Epub 2020 Mar 23. PMID 32202965
- [Background] Ibrahim LA, Tawfik MN, Naeem FMA. Evaluation of The Periapical Healing Following Pulp Revascularization Using Injectable PRF VS nonsurgical Root Canal Treatment in Mature Permanent Teeth with periapical periodontitis. A Clinical Study. Egypt Dent J. 2021;67(3):2663-2672